CLINICAL TRIAL: NCT00286949
Title: Atomoxetine for the Treatment of Executive Dysfunction in Patients With Parkinson's Disease: A Pilot Open-label Study
Brief Title: Treatment of Executive Dysfunction in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIRB#20040223; B4Z-US-X029 (Other: Eli Lilly Investigator-Initiated Grants Program)
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; executive dysfunction; impairment; motor skills; cognitive
MeSH Terms: conditions — Parkinson Disease | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atomoxetine (Strattera) (Other): Open-Label Uncontrolled Active Drug Intervention, No comparator
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — Open Label uncontrolled active Drug intervention
  Other Names: Strattera (Brand Name)

SUMMARY:
Atomoxetine (Strattera) is a drug that is currently approved for treatment of attention deficit hyperactivity disorder (ADHD) in children and adults. Atomoxetine works to enhance levels of brain chemicals that may be affected in people with executive dysfunction, (difficulties with organization, task completion, and priority setting). Thus, atomoxetine has the potential to improve executive dysfunction in people with Parkinson's disease (PD).

The goal of this study is to provide preliminary data on the effectiveness and tolerability of atomoxetine for the treatment of executive dysfunction in patients with PD.

DETAILED DESCRIPTION:
Parkinson's disease (PD), while defined by its motor abnormalities and associated dopaminergic loss, is invariably accompanied by cognitive impairment. Early in the disease course, the deficits are characterized by executive dysfunction with difficulties on tasks that involve information processing, attention, sorting, planning, set-shifting, and working memory and are subserved by neural connections with prefrontal brain regions. There has been little effort to identify treatments for these PD-related cognitive impairments, despite their disabling and distressing effects. Accordingly, the goal of this proposal is to conduct a small pilot study to determine the effectiveness and tolerability of atomoxetine, a selective norepinephrine reuptake inhibitor, for the treatment of executive dysfunction in patients with PD.

Atomoxetine (Strattera) is currently approved by the FDA for treatment of attention deficit hyperactivity disorder (ADHD) in children and adults. Atomoxetine enhances dopaminergic and noradrenergic transmission in frontal regions that are also implicated in executive dysfunction and thus has the potential to improve executive dysfunction in PD as well as other neurological conditions. Results of the study will be used to develop a larger placebo-controlled trial of atomoxetine, if appropriate, as well as inform the design of other clinical trials on potential treatments for cognitive dysfunction in PD.

The overall hypothesis is that atomoxetine will be an effective and safe treatment for executive dysfunction in PD.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with idiopathic Parkinson's Disease, as defined by United Kingdom (UK) Brain Bank Criteria.
2. Adults, ages 21 to 65 years old.
3. Clinically significant executive dysfunction, as defined by the reported presence of problems with disorganization, distractibility, task completion, planning or problem solving that represents a decline from premorbid (pre-PD) status and is confirmed by the patient's informant.
4. Mini-Mental State Exam (MMSE) score > 26.
5. Absence of Dementia due to Parkinson's Disease, as defined by Diagnostic and Statistical Manual-IVth edition-Text revision (DSM-IV-TR).
6. Clinical Dementia Rating (CDR) Scale score < 1.
7. Functional Assessment Staging (FAST) score < 4.
8. Hamilton Depression Rating Scale (HDRS) Score < 11.
9. Able to provide informed consent and participate in follow-up visits during the 8-week study duration.
10. Availability of informant who knows the patient well and is willing to provide collateral information on the patient's clinical status and response to treatment.
11. On stable antiparkinsonian therapy for 3 months.
12. Any stage of PD severity, e.g., Hoehn and Yahr stage I-V, but must be able to participate in testing battery and be capable of independent function so as to manifest executive dysfunction.
13. Stable medical health with stable medication regimen for 3 months.
14. If history of major depression or anxiety disorder, must have stable symptoms and be on stable therapy for 3 months.
15. For women of childbearing potential, negative pregnancy test and reliable use of contraception.

Exclusion Criteria:

1. Prior exposure to atomoxetine within the last 6 months.
2. Current problems with urinary hesitancy or urinary retention.
3. Uncontrolled hypertension or tachycardia.
4. Narrow angle glaucoma.
5. Current presence of hallucinations without insight or uncontrolled delusions (patients with benign visual hallucinations of any sensory modality with insight, e.g., passage or presence hallucinations, or controlled stable delusions will be enrolled).
6. Illicit substance use or alcohol abuse or dependence within the last 6 months.
7. Current symptomatic Major Depressive Disorder or Anxiety Disorder that warrants additional treatment, as assessed on clinical interview, or 21-item Hamilton Depression Scale > 10.
8. For women, current pregnancy or nursing.
9. Current use of potent CYP2D6 inhibitors, e.g., paroxetine, fluoxetine, quinidine.
10. Current use of stimulant or wakefulness therapy, e.g., methylphenidate or modafinil.
11. Current hepatic dysfunction, defined as values of two times or greater than the upper limit of normal on the aspartate aminotransferase (AST) or alanine aminotransferase (ALT) hepatic enzymes or any disorder affecting the liver that in the opinion of the enrolling investigator would interfere with hepatic metabolism of the medication or interfere with the participant's ability to complete the study.
12. Current use of monoamine oxidase inhibitors that are typically used for treatment of depression (isocarboxazid, phenelzine, and tranylcypromine).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-01-06 (Actual); Primary Completion 2008-06-30 (Actual); Study Completion 2008-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Marsh, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marsh L, Biglan K, Gerstenhaber M, Williams JR. Atomoxetine for the treatment of executive dysfunction in Parkinson's disease: a pilot open-label study. Mov Disord. 2009 Jan 30;24(2):277-82. doi: 10.1002/mds.22307. PMID 19025777

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parkinson's disease (PD) outpatients (recruited 2005-2008 via Johns Hopkins clinics and community) had clinically significant Executive Dysfunction, defined as moderately severe problems with disorganization, distractibility, task completion, planning or problem solving that impaired function, were a decline from pre-PD, and verified by informant.
Pre-assignment Details: All enrolled subjects were assigned to and received open label atomoxetine.
Groups:
- Atomoxetine Open Label: This open-label, uncontrolled, single arm, flexible dose trial consisted of atomoxetine (Strattera) in 25 mg capsules initiated at 25 mg/day in the morning (Week 1) and advancing to 50mg/at (weeks 2-4), 75 mg/day (Week 5), and 100 mg/day (Weeks 6-8). Dose reductions were allowed to a minimum of 2.5 mg/day for intolerance.
Period: Overall Study
Arm/Group | Atomoxetine Open Label
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Atomoxetine: Atomoxetine (Strattera): Open label, no comparator
Arm/Group | Atomoxetine
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression of Change-Clinician Rated Score (CGIC-C)
Description: CGIC-C score is a clinician's rating of change (improvement or worsening) over the course of the trial in an individual's symptoms and their global impact on function and clinical status, i.e., the global impact of the intervention that the patient is better, unchanged, or worse). Scale ranges1 to 7 which equates to from very much worse to very much improved.
  The CGIC-C score is not an appropriate baseline measure since it represents change after initiating an intervention. In addition, a baseline Clinical Global Impression of Severity-Clinician Rated Score (CGIS-C) is not appropriate to compare to CGIC-C, as a patient with severe disease might show clinically meaningful improvement (i.e., very much improved) from an intervention while still being severely affected on the CGIS-C score; by contrast, a patient with mild CGIS-C could have minimal or no change on the CGIC-C score. This study was not designed to assess the influence of disease severity on the primary outcome (CGIC-C).
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Atomoxetine Open Label: Active open label drug, no comparator; Atomoxetine (Strattera)
Arm/Group | Atomoxetine Open Label
Number analyzed (Participants) | 12
Participants
  Very Much Improved | 3
  Much Improved | 6
  Minimally Improved | 1
  No Change | 2
  Minimally Worse | 0
  Much Worse | 0
  Very Much Worse | 0

2. Primary Outcome: Connors Adult Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale-Long Form (CAARS-L) Inattention/Memory Subscale
Description: The CAARS-L Inattention/Memory subscale, a primary self-rated outcome measure in this study, measures the frequency of behaviors associated with executive dysfunction, such as task incompletion, disorganization, distractibility, and difficulty planning, multi-tasking, and initiating tasks. CAARS-L scores are depicted as group Mean (SD) T scores, derived from comparison to CAARS norms based on gender and age in a normative sample. Similar to the FrSBE, higher T-scores are associated with greater symptom severity and T-scores above 65 represent symptoms of clinical significance.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine (Strattera)
Number analyzed (Participants) | 12
units on a scale
  Baseline Visit | 60 (10)
  Final Visit (8 weeks) | 52 (10)

3. Primary Outcome: Frontal Systems Behavioral Scale (FrSBe) Executive Function Subscore
Description: Frontal Systems Behavioral Scale (FrSBe) Executive Function subscore is on of the 3 subscales of the FrSBE, a scale designed to identify and quantify behavioral problems associated with frontal lobe dysfunction. The other subscales are Apathy and Disinhibition. Each item is rated on a 5-point Likert scale. Totals are generated for each subscale and normative data is referenced (based on patient gender, age and education) and standardized T-scores are determined). For all FrSBe scales, T scores ≥ 65 are considered clinically significant and scores of 60 to 64 represent likely borderline impairment.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Atomoxetine: Active open label drug, no comparator
  Atomoxetine (Strattera)
Arm/Group | Atomoxetine
Number analyzed (Participants) | 12
T-score
  Baseline Visit | 67 (11)
  Final Visit | 58 (15)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Vital signs, spontaneously reported adverse events (AEs), Udvalg for Kliniske Undersogelser (UKU) AE checklist,Unified Parkinson's Disease RatingScale (UPDRS)-Activities of Daily Living, Motor, and Complications of Therapy subscales,Hoehn and Yahr Stage,changes from baseline labor tests, and cardiovascular effects
Groups:
- Atomoxetine: Open label, no comparator
  Atomoxetine (Strattera)
Arm/Group | Atomoxetine
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=12)
Hypomania (Psychiatric disorders) | 1 (1) — One subject developed hypomania on atomoxetine 75 mg/day that remitted with reduction to 25 mg/day.
Reduced Sleep (Nervous system disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 5 (5)
Nausea/vomiting (Gastrointestinal disorders) | 3 (3)
Confusion (Nervous system disorders) | 3 (3)
Slowed movements (Nervous system disorders) | 3 (3)
Diaphoresis (Skin and subcutaneous tissue disorders) | 3 (3)
Fatigue (General disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2)
increased dream activity (Nervous system disorders) | 2 (2)
Rigidity (Nervous system disorders) | 2 (2)
Hyperkinetic movements (Nervous system disorders) | 2 (2)
paresthesias (Nervous system disorders) | 2 (2)
Headaches (Nervous system disorders) | 2 (2)
Dry mouth (General disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Weight gain (General disorders) | 2 (2)
Dysmenorrhea (Reproductive system and breast disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Data interpretation limited by open-label uncontrolled design, small sample size, subjects young (< age 65 years); multiple comparisons, intersubject variability, possible inclusion bias, ceiling and practice effects for neuropsychological data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No